CLINICAL TRIAL: NCT00351416
Title: Letrozole Treatment in Normal and GnRH Deficient Women
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Janet E. Hall, MD, Associate Physician, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 2003-P-001895; Sundry Department Fund (Other: MGH-REU Department Fund)
Record Dates: First submitted 2006-07-10; First posted 2006-07-12 (Estimated); Results first posted 2017-04-27 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2017-06

CONDITIONS: Healthy Volunteers
Keywords: GnRH deficiency; GnRH antagonist; Letrozole; GnRH; FSH; LH; Inhibins
MeSH Terms: interventions — Letrozole; Aromatase Inhibitors; LHRH, Ac-Nal(1)-Cpa(2)-Trp(3)-Arg(6)-Ala(10)-

STUDY DESIGN:
Intervention Model Description: This is a physiologic study designed to investigate the relative roles of estradiol and inhibin A or inhibin B in the control of FSH secretion during normal menstrual cycles using an aromatase inhibitor. Subjects serve as their own control with no intervention in cycle 1 and letrozole administration in cycle 2. Subjects are studied in the early follicular phase or the late follicular phase.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Aromatase inhibitor EFP (Experimental): Letrozole administration (20 mg) on day 2-4 (EFP; early follicular phase) of cycle 2 and
  Nal-Glu GnRH antagonist used to estimate the overall amount of GnRH secreted.
  Interventions: Drug: Letrozole; Drug: NAL-GLU GnRH antagonist
- Aromatase inhibitor LFP (Experimental): Letrozole administration (20 mg daily x 2) at follicle size of > 16 mm (LFP; late follicular phase) in cycle 2.
  Nal-Glu GnRH antagonist used to estimate the overall amount of GnRH secreted.
  Interventions: Drug: Letrozole; Drug: NAL-GLU GnRH antagonist

INTERVENTIONS:
Drug: Letrozole — Letrozole 20 mg orally one time
  Other Names: aromatase inhibitor; Femara
Drug: NAL-GLU GnRH antagonist — 5 mcg/kg of the NAL-GLU GnRH antagonist subcutaneously
  Other Names: GnRH antagonist

SUMMARY:
This research study involves the use of the drugs Letrozole, GnRH, and NAL-GLU GnRH antagonist. Letrozole is a drug that is approved by the U.S. Food and Drug Administration (FDA) for use in breast cancer treatment that has been found to block the formation of estrogen. The NAL-GLU GnRH antagonist is a drug that temporarily blocks the action of GnRH. GnRH is a hormone that the body makes that stimulates other hormones that then control the function of the ovary.

The purpose is to study the effects of the administration of letrozole in women with GnRH deficiency at the same time that they receive gonadotropin-releasing hormone (GnRH). In addition, administration of letrozole and NAL-GLU GnRH antagonist in healthy women with normal menstrual cycles will be done to evaluate the role of estrogen in the control of the hormone FSH, or Follicle Stimulating Hormone, in the female reproductive cycle. A better understanding of FSH control may help in the development of new treatments for women with difficulty conceiving.

DETAILED DESCRIPTION:
The negative feedback control of FSH is crucial for the precise regulation of follicular development in the female. An important component of this feedback is exerted by estrogen. Letrozole will be used to block aromatase and therefore estradiol production in normal and GnRH deficient females. These studies will dissect the relative roles of estradiol and inhibin on FSH secretion at the pituitary and hypothalamus.

The aromatase inhibitors block aromatization of androgens to estrogens, allowing us to examine the relative contribution of estradiol and the inhibins to FSH regulation. The use of a submaximal dose of a GnRH antagonist will allow us to estimate the overall amount of GnRH secreted (hypothalamic contribution) with and without aromatase inhibition.

A more thorough understanding of estrogen and inhibin feedback on FSH will improve our understanding of the failure of follicle development in subsets of patients with infertility, such as polycystic ovary syndrome, in which FSH levels are normal but follicles fail to develop. Study of FSH control will also help us understand the failure of negative feedback on FSH, which can result in multiple follicular development and multiple gestation and its associated costs and risks. Thus, these studies may afford new therapeutic options for conception in infertile patients while simultaneously providing new methods to avoid the risks of multiple gestations.

ELIGIBILITY:
Inclusion Criteria:

Healthy Normal Subjects will meet the following criteria:

* 18 to 35 years of age
* good general health
* on no medications including any hormonal drug products for at least 3 months before the study
* regular menstrual cycles every 25-35 days with ovulation documented by a luteal phase progesterone > 3 ng/ml
* no evidence of androgen excess
* normal TSH, prolactin and hemoglobin
* use of double-barrier contraception, permanent sterilization or abstinence during the cycle of study.
* Negative pregnancy test (serum) at the beginning of each cycle of study
* Normal Liver Function Test

Exclusion Criteria:

* History of liver and/or kidney disease
* Substance or alcohol abuse
* Hormone dependent neoplasia including breast cancer
* Women who are trying to become pregnant

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 15 (Actual)
Dates: Start 2004-01-21 (Actual); Primary Completion 2009-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet E Hall, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Reproductive Endocrine Unit, Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Once published, de-identified individual level data will be shared upon request to the PI.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Four subjects did not meet inclusion criteria (2 had increased prolactin, 2 had abnormal cycles) and were excluded after screening and before assignment to treatment.
Groups:
- Aromatase Inhibitor EFP: Letrozole administration (20 mg) on day 2-4 (EFP; early follicular phase) of cycle 2 and
  Nal-Glu GnRH antagonist used to estimate the overall amount of GnRH secreted.
  Letrozole: Letrozole 20 mg orally one time
  NAL-GLU GnRH antagonist: 5 mcg/kg of the NAL-GLU GnRH antagonist subcutaneously
- Aromatase Inhibitor LFP: Letrozole administration (20 mg daily x 2) at follicle size of > 16 mm (LFP; late follicular phase) in cycle 2.
  Nal-Glu GnRH antagonist used to estimate the overall amount of GnRH secreted.
  Letrozole: Letrozole 20 mg orally one time
  NAL-GLU GnRH antagonist: 5 mcg/kg of the NAL-GLU GnRH antagonist subcutaneously
Period: Overall Study
Arm/Group | Aromatase Inhibitor EFP | Aromatase Inhibitor LFP
Started | 6 | 9
Completed | 6 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aromatase Inhibitor EFP | Aromatase Inhibitor LFP | Total
Number analyzed (Participants) | 6 | 9 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.2 (5) | 28.5 (4.2) | 27.9 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 5 | 8 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 4 | 8 | 12
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 9 | 15

OUTCOME MEASURES:

1. Primary Outcome: FSH Level
Description: Difference in FSH peak following letrozole administration compared with control cycle
Time Frame: EFP: average of menstrual cycle day 6 in the EFP; LFP: average of 2 days after follicle size of 16 mm
Measure: Mean (Standard Error); unit: IU/L
Arm/Group | Aromatase Inhibitor EFP | Aromatase Inhibitor LFP
Number analyzed (Participants) | 6 | 9
IU/L | 7.25 (2.42) | 8.71 (1.58)

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Aromatase Inhibitor EFP | Aromatase Inhibitor LFP
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No